CLINICAL TRIAL: NCT00675766
Title: Aging & HIV/AIDS Neurocognitive Sequelae and Functional Consequences
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: AGCG-012-04F
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: HIV-positive adults 50 and older/ HIV-positive adults 18-40 years old
- Group 2: HIV-negative controls 50 and older / HIV-negative controls 18-40 years old
- Group 3: HIV-negative controls 50 and older / HIV-negative controls 18-40 years old
- Group 4: HIV-negative controls 18-40 years old

SUMMARY:
While the numbers of HIV infected veterans under the age of 50 are declining, the percentage of HIV infected veterans over the age of 50 is increasing with the largest percentage increases in the 50-59 age group and the 70+ age group. With increasing incidence rates of new cases among individuals over 50 years of age and the longer life expectancies of the current HIV-infected population, it becomes increasingly important to better understand the impact of the aging process on the clinical and behavioral manifestations of HIV/AIDS.

The project seeks to determine the effect of age on neuropsychological performance in HIV+ persons. This objective seeks to determine the degree to which older age represents an independent risk factor for neuropsychological impairment in HIV infected persons, with a particular emphasis on those cognitive processes that are preferentially impacted by both the normal aging process as well as HIV infection. Additionally, another aim of the study is to determine the impact of neuropsychological decline on everyday functional abilities among older vs. younger HIV+ adults. This objective seeks to determine the effects of advancing age and neuropsychological impairment on the ability of HIV+ persons to discharge more demanding requirements of independent living (e.g., driving, financial management, medication adherence). The project will last for a duration of 5 years.

DETAILED DESCRIPTION:
Over the past several years the HIV epidemic has changed from a disease primarily of younger, gay/bisexual, Caucasian men to one increasingly affecting people of color, women, and, of specific relevance to this application, the older adult. Indeed, the number of AIDS cases in individuals over the age of 50 has more than tripled over the last several years, with the CDC now estimating that in the United States 15% of all patients with AIDS are over age 50.1 There is reason to believe that the incidence, clinical manifestations and course of HIV-associated CNS dysfunction may differ as a function of age. Since the mid 1980's VA has been at the vanguard of institutions engaged in research and clinical care of HIV-infected adults. With specific regard to the issue of aging and HIV, HIV-infected veterans have tended to be significantly older than patients drawn from the general community. For example, at the West Los Angeles VA 303 of the 583 (52%) HIV-infected patients being followed by the Infectious Disease clinic are over the age of 50. Across the entire VA system, there are nearly twice as many HIV infected veterans over the age of 70 than under 30 years of age. 2 Yet, the vast majority of research conducted to date has been on younger adults - the degree to which such data will generalize to the older veteran population is unclear. Also unclear is whether advancing age confers an independent risk for cognitive impairment in HIV-infected persons. Additionally, the functional impact (i.e., impact on daily functioning such as driving ability, financial management, or medication adherence) of cognitive impairment in this group remains unknown. Exploratory studies performed in the applicants' laboratory have provided preliminary support for the hypothesis that advancing age will potentiate the deleterious neurocognitive effects of HIV infection. Given the "graying" of the HIV epidemic, particularly among the veteran population, research examining neurocognition among older HIV-infected veterans as well as the functional "real world" impact of such deficits is of great relevance to the VA mission. The results from this study could provide important insights into interactions of age and HIV disease, and will identify targets for intervention in advance of the burgeoning population of older infected persons.

SPECIFIC OBJECTIVES AND HYPOTHESES

Objective 1. To Determine the Effect of Age on Neuropsychological Performance in HIV+ Persons This objective seeks to determine the degree to which older age represents an independent risk factor for neuropsychological impairment in HIV infected persons, with a particular emphasis on those cognitive processes that are preferentially impacted by both the normal aging process as well as HIV infection.

Hypothesis 1.1 Controlling for potential confounding factors such as substance use and length of infection, there will be an interaction between effects of age and HIV serostatus on neuropsychological performance, and this will be evident both cross-sectionally and longitudinally. Specifically, we expect to find that older HIV+ individuals will exhibit greater rates of neuropsychological impairment (using age-corrected test norms) than younger HIV+ persons. Neurocognitive functions subserved by frontal-subcortical systems that are sensitive to the effects of both aging and HIV infection (learning, motor and psychomotor speed, executive function) will be disproportionately affected among the older HIV+ participants. While the synergistic effects of HIV and age will be evident on a cross sectional basis, they will be most pronounced when examined longitudinally over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in the study, participants must be between the ages of 18-40 years (younger groups) or > 50 years (older groups); our goal is to recruit at least 50% of older HIV+ participants who are > 60 years old.
* Eligible participants must have documented presence or absence of HIV infection (depending on their group assignment), based on serologic testing for HIV antibody (screening ELISA, confirmed by Western blot if positive).
* The documentation of HIV status will be obtained once informed consent has been established.

Exclusion Criteria:

* CNS infection other than HIV (no opportunistic CNS disease)
* CNS neoplasm, neurosyphilis
* traumatic brain injury with loss of consciousness greater than 30 minutes
* current diagnosis of seizure disorder, current psychotic spectrum disorders (e.g., schizophrenia, bipolar disorder)
* history of drug or alcohol abuse or dependence within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To be enrolled in the study, participants must be between the ages of 18-40 years (younger groups) or 50 years old and older (older groups). The study population will consist of an ethnically diverse sample of approximately 1/3 Caucasian, 1/3 African American and 1/3 Hispanic. Approximately, 25% of participants will be female. The population will consist of veterans with additional recruitment from the community in order to meet project goals.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2005-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hinkin, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

REFERENCES:
- [Derived] Foley JM, Gooding AL, Thames AD, Ettenhofer ML, Kim MS, Castellon SA, Marcotte TD, Sadek JR, Heaton RK, van Gorp WG, Hinkin CH. Visuospatial and Attentional Abilities Predict Driving Simulator Performance Among Older HIV-infected Adults. Am J Alzheimers Dis Other Demen. 2013 Mar;28(2):185-94. doi: 10.1177/1533317512473192. Epub 2013 Jan 11. PMID 23314403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from September 2005 to September 2010. The population consisted of young (40 years or less) and old (50 years or more) Human Immunodeficiency Virus infected and non-infected veterans within the Greater Los Angeles VA Healthcare System with additional recruitment from the Los Angeles community in order to meet project goals.
Pre-assignment Details: Recruited subjects who meet any of the following criteria were excluded prior to group assignment: Brain infection other than HIV; Brain neoplasm; neurosyphilis; traumatic brain injury with L.O.C>30 mins; current diagnosis of seizure disorder; current psychotic spectrum disorders; history of drug or alcohol abuse or dependence within the past year.
Groups:
- Group 1: HIV-positive adults 50 and older
- Group 2: HIV-positive adults 18-40 years old
- Group 3: HIV-negative controls 50 and older
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 106 | 30 | 50 | 37
Year 2 | 105 | 28 | 34 | 20
Year 3 | 100 | 25 | 29 | 11
Completed | 100 | 25 | 29 | 11
Not Completed | 6 | 5 | 21 | 26
Not completed — Lost to Follow-up | 6 | 5 | 21 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 106 | 30 | 50 | 37 | 223
Age, Customized [Number; unit: participants]
  Between 18 and 40 years old | 0 | 30 | 0 | 37 | 67
  50 years and older | 106 | 0 | 50 | 0 | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 6 | 32 | 17 | 73
  Male | 88 | 24 | 18 | 20 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 0 | 4
  Asian | 1 | 1 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 59 | 12 | 36 | 16 | 123
  White | 43 | 15 | 9 | 12 | 79
  More than one race | 1 | 2 | 2 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 106 | 30 | 50 | 37 | 223

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Status (i.e., Cognitive Functioning)
Description: Neurocognitive functions refer to cognitive abilities, namely learning/memory, motor speed, psychomotor speed, language, attention, visuospatial abilities, & executive function. They are measured using standard clinical neuropsychological test battery that included: HVLT, BVMT-R, Trails A & B, WCST-64, WAIS-Symbol Search/Digit Coding/Letter-Number Sequencing/Block Design, FAS, & Animals. Subgroups of these tasks were combined to create composite scores indicating participants' score on each cognitive domains. To make these cognitive domain composite scores, each participant's raw score on each of these tests was converted into a within-sample standardized score (i.e., z-score), which are normally distributed with a mean of 0 & SD of 1. Then, these standardized scores were summed to create composite scores for each cognitive domain and then averaged to create a global neuropsychological function composite score. A positive composite score represents a better outcome for all variables.
Time Frame: Baseline (Year 1) and 1-year follow-up (Year 2)
Population: HIV+ and HIV negative men who were evaluated BOTH at baseline and Year 2. Those participants who were evaluated at Baseline but not at Year 2 were excluded from analyses.
Measure: Mean (Standard Error); unit: z-score composites of cognitive domains
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 67 | 16 | 15 | 5
z-score composites of cognitive domains
  Baseline z-score global neurocognitive composite | 0.008 (.066) | .484 (.134) | -.084 (.157) | -.482 (.301)
  Year 2 z-score global neurocognitive composite | -.091 (.066) | .517 (.134) | -.036 (.157) | .397 (.300)
  Baseline z-score for language | 0.056 (0.762) | 0.468 (0.520) | -.075 (.480) | -.112 (.835)
  Year 2 z-score for language | 0.014 (.840) | .413 (.773) | -.088 (.680) | .385 (.605)
  Baseline z-score for learning/memory | -.034 (.875) | .540 (.618) | -.287 (.552) | .277 (1.338)
  Year 2 z-score for learning/memory | -.145 (.832) | .493 (.689) | -.126 (.884) | .360 (.630)
  Baseline z-score for attention | .035 (.870) | .215 (.681) | .070 (.816) | -.190 (1.396)
  Year 2 z-score for attention | -.026 (.816) | .366 (.654) | -.199 (.863) | .706 (.435)
  Baseline z-score for processing speed | -.043 (.729) | .602 (.469) | -.301 (.552) | -.241 (.831)
  Year 2 z-score for processing speed | -.167 (.726) | .600 (.761) | -.422 (.699) | .586 (.496)
  Baseline z-score for executive function | -.047 (.417) | .331 (.397) | -.221 (.564) | -.318 (.832)
  Year 2 z-score for executive function | -.052 (.843) | .292 (.360) | -.070 (.484) | -.029 (.086)
  Baseline z-score for visuospatial function | -.020 (.923) | .801 (1.013) | -.163 (.788) | .450 (.975)
  Year 2 z-score for visuospatial function | -.144 (.892) | .859 (.820) | -.153 (.927) | .821 (.485)
  Baseline z-score for motor speed | .009 (.862) | .516 (.632) | -.356 (.993) | -.091 (.836)
  Year 2 z-score for motor speed | .093 (.817) | -.515 (.411) | .177 (.696) | -.446 (.371)
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with overall neurocognitive performance at baseline and follow-up, computed as z-scored derived composite score of 14 individual neuropsychological measures assessing attention, processing speed, visuospatial skills, language, memory, executive function and motor skills, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p = 0.001, Repeated Measures ANOVA; Range of z-scores at baseline: -1.69 to 1.38. Range of z-scores at Year 1 follow-up: -1.28 to 1.36
Statistical Analysis 2: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with processing speed at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing speed of cognitive information processing, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p < 0.005, Repeated Measures ANOVA; Range of z-scores at baseline: -2.96 to 1.89. Range of z-scores at Year 1 follow-up: -1.89 to 1.77
Statistical Analysis 3: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with attention at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing attentional abilities, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p < 0.01, Repeated Measures ANOVA; Range of z-scores at baseline: -2.30 to 2.44. Range of z-scores at Year 1 follow-up: -1.82 to 2.00
Statistical Analysis 4: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with executive function at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing working memory, set shifting, mental flexibility and problem solving, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p < 0.07, Repeated Measures ANOVA; Range of z-scores at baseline: -1.76 to 0.95. Range of z-scores at Year 1 follow-up: -1.18 to 0.84
Statistical Analysis 5: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with language at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing verbal fluency and naming skills, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p = 0.09, Repeated Measures ANOVA; Range of z-scores at baseline: -2.30 to 1.94. Range of z-scores at Year 1 follow-up: -1.83 to 2.11
Statistical Analysis 6: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with memory at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing verbal and nonverbal learning and memory, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p = .72, Repeated Measures ANOVA; Range of z-scores at baseline: -2.00 to 1.68. Range of z-scores at Year 1 follow-up: -2.33 to 1.90
Statistical Analysis 7: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with visuospatial skills at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing visuospatial and visuoconstructional abilities, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p = 0.65, Repeated Measures ANOVA; Range of z-scores at baseline: -2.04 to 2.51. Range of z-scores at Year 1 follow-up: -2.21 to 2.24
Statistical Analysis 8: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Repeated Measures ANOVA with motor skills at baseline and follow-up, computed as z-scored derived composite score of multiple neuropsychological measures assessing fine motor speed and dexterity, across time as the within-group factor and HIV serostatus and age group as between-group factors; Test type: Superiority or Other; p = 0.79, Repeated Measures ANOVA; Range of z-scores at baseline: -4.04 to 1.33. Range of z-scores at Year 1 follow-up: -1.24 to 2.37
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Fisher's exact test compared the frequency of older and younger HIV+ adults who converted from neurocognitively intact to neurocognitively impaired on memory over a one year time period. We hypothesized that the older group would exhibit a greater proportion of individuals who declined during this interim; Test type: Superiority or Other; p = .044, Fisher Exact; One-sided Fisher's exact test with 1 degree of freedom

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 4 years after each subject's baseline visit.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/30 | 0/50 | 0/37
Other Adverse Events (participants affected / at risk) | 0/106 | 0/30 | 0/50 | 0/37

LIMITATIONS AND CAVEATS:
Large number of subjects who were lost to follow up (i.e moved from community, did not answer follow up calls to schedule visits) resulted in a reduced sample size of subjects who completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No